CLINICAL TRIAL: NCT01470768
Title: Evaluation of Fatty Acid Levels and Growth in Infants Fed Amino Acid Based Formulas
Brief Title: Evaluation of Fatty Acid Levels and Growth in Infants Fed Amino Acid Based (AA) Formulas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor cancelled study
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 6005
Record Dates: First submitted 2011-10-26; First posted 2011-11-11 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Cow's Milk Allergy; Intolerance to Extensively Hydrolyzed Formulas; Intolerance to Breast Milk
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 - AA Formula with DHA and ARA (Other): Marketed AA formula with Docosahexanoic Acid (DHA) and Arachidonic Acid (ARA)
  Interventions: Other: Amino Acid-based Formula with high DHA and ARA
- Arm 2 - AA Formula with alternative levels of DHA and ARA (Other)
  Interventions: Other: Amino Acid-based Formula with lower DHA and ARA

INTERVENTIONS:
Other: Amino Acid-based Formula with high DHA and ARA
  Arms: Arm 1 - AA Formula with DHA and ARA
Other: Amino Acid-based Formula with lower DHA and ARA
  Arms: Arm 2 - AA Formula with alternative levels of DHA and ARA

SUMMARY:
This clinical trial will compare the amount of fatty acids in whole blood of babies fed one of two study formulas for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 6 months of age inclusive
* Born at ≥ 37 weeks gestation
* Birth weight of 2500 g (5 lb 8 oz) or more
* Infants suspected to be cow's milk allergic and who do not tolerate extensively hydrolyzed formula OR infants intolerant to breast milk
* Infants with symptoms suggestive of cow's milk allergy
* Signed Informed Consent

Exclusion Criteria:

* Infants who for whatever reasons were not discharged home as per routine
* Infants with metabolic illness requiring a special formula
* Infants fed with nasogastric tube

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Level of fatty acids in whole blood of infants | 4 months

SECONDARY OUTCOMES:
body weight | 4 months
Occurrence of allergic manifestations | 4 months
Occurrence of adverse events | 4 months
Incidence of gas | 4 months
Incidence of fussiness | 4 months
Stool characteristics | 4 months
Body length | 4 months
Head Circumference | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Thapar, M.D., Principal Investigator — UCL Institute of Child Health and Great Ormond Street Hospital
Locations (1):
- Great Ormand Street Hospital and Institute of Child Health, London, United Kingdon, United Kingdom

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765